CLINICAL TRIAL: NCT06076005
Title: Demographic, Clinical, Histological and Molecular Characteristics of Advanced LUNG CANCER at the tIme of Diagnosis in a Large Italian Cohort, an Observational Cohort Study: Lung Cancer ID Study
Brief Title: Characteristics of Advanced LUNG CANCER at the tIme of Diagnosis in a Large Italian Cohor
Acronym: LUNG-CANCER
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5937
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer Stage IV
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Advanced lung cancer patients' group — Evaluation of the demographic, clinical, histological and molecular characteristics of advanced lung cancer at the time of Diagnosis

SUMMARY:
The distribution of demographic, clinical, radiological, pathological and molecular characteristics of lung cancer at the time of diagnosis, as well as preferential association between elements of those domains, have not been specifically studied in Italy. The aim of the present project is to assess, in a systematic fashion, the demographic, clinical, radiological, pathological and molecular characteristics of advanced lung cancer at the time of diagnosis in a large Italian cohort of consecutive patients referred to two tertiary referral centers.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Suspicion of lung cancer based on imaging (CT and/or PET/CT)
* Indication to a biopsy for diagnosis, staging and/or molecular profiling

Exclusion Criteria:

* Inability or unwillingness to provide a written informed consent
* ECOG performance status (>3) which makes a tissue diagnosis unfeasible
* ASA 4 status
* TNM Stage I-III

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive, treatment-naïve, patients with clinical and radiological suspicion of advanced lung cancer referred for the initial diagnosis/staging/molecular profiling.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Distribution of histologic subtypes | 24 months
  The investigators will assess the prevalence of histologic subtypes in patients with advanced lung cancer

SECONDARY OUTCOMES:
Distribution of histologic subtypes according to clinical and radiological characteristics | 24 months
  The investigators will assess the prevalence of different histologic subtypes according to clinical and imaging characteristics
Molecular profiling | 24 months
  Prevalence of individual molecular markers in patients with advanced non-squamous non-small cell lung cancer histology
Time to diagnosis | 24 months
  Time lag between onset of symptoms (if any) and invasive testing

CONTACTS AND LOCATIONS:
Overall Officials: Rocco Trisolini, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (3):
- Italy (3):
  - Interventional Pulmonology Division - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Medical Oncology Division - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma

IPD SHARING:
Plan to Share IPD: Undecided
The investigators will decide how to share the data at the end of the study upon reasonable request to be addressed to the principal investigator.